CLINICAL TRIAL: NCT05550441
Title: Effect of Sodium-dependent Glucose Transporters 2 Inhibitor Dapagliflozin on Ventricular Arrhythmia in Patients With Heart Failure.
Brief Title: Effect of Dapagliflozin on VT in Patients With Heart Failure.
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, Shuxian Zhou, Clinical Professor, Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2020-KY-129
Record Dates: First submitted 2022-06-15; First posted 2022-09-22 (Actual); Last update posted 2022-09-22 (Actual); Status verified 2022-09

CONDITIONS: Heart Failure
Keywords: heart failure; dapagliflozin; ventricular arrhythmia; clinical randomized controlled trial
MeSH Terms: conditions — Heart Failure | interventions — dapagliflozin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Placebo group (Placebo Comparator)
  Interventions: Drug: Placebo
- Dapagliflozin group (Experimental)
  Interventions: Drug: Dapagliflozin

INTERVENTIONS:
Drug: Dapagliflozin — The experimental group received dapagliflozin (10 mg qd) for 1 year.
  Arms: Dapagliflozin group
Drug: Placebo — The Placebo group received placebo for 1 year.
  Arms: Placebo group

SUMMARY:
This project plans to design a randomized controlled clinical trial to evaluate the effect of dapagliflozin on ventricular arrhythmia in the participants with heart failure with reduced ejection fraction after ICD implantation by collecting and analyzing the data of ECG, cardiac ultrasound and ICD programming. This project will explore the anti-ventricular arrhythmia effect of dapagliflozin in HFrEF patients.

DETAILED DESCRIPTION:
This is a single-center, randomized, controlled, double-blind study in Chinese heart failure participants with ICD implantation. This trial aims to investigate the effect of dapagliflozin on ventricular arrhythmias in participants with HFrEF. This trial includes a screening period, a treatment period and a follow-up period. Total duration of each subject's participation in the trial is approximately 1 year. During the screening period, 120 participants with HFrEF with ICD implanted in the investigator's department were recruited. The participants should sign the informed consent and be randomly divided into 2 groups. All participants will receive the best anti-heart failure treatment for 6 months before enrollment, including ACEI/ARB/ARNI, β-blockers, spironolactone, diuretics, and digitalis. One group was randomized to receive dapagliflozin (10 mg qd) and another group received place. Participants were then enrolled in a 1-year clinical trial and investigators will record the participants' QT interval, QTc interval, frequency and mode of ICD electrical therapy, cardiac function, symptoms, signs and other indicators before and after treatment to evaluate the occurrence of ventricular arrhythmia.

ELIGIBILITY:
Inclusion Criteria:

patients received ICD therapy with HFrEF, including: ischemic cardiomyopathy, non-ischemic cardiomyopathy, LVEF ≤35% and optimized anti-HF therapy for at least 6 months.

Exclusion Criteria:

1. Type 1 diabetes or a history of repeated diabetic ketoacidosis.
2. Those who strictly restrict carbohydrate intake.
3. Genital infection.
4. Low blood pressure.
5. SGLT2i allergy.
6. Severe renal impairment or end-stage renal disease (eGFR<30ml/(min•1.73m^2)) or dialysis.
7. The water-electrolyte and acid-base balance disorders have not been corrected.
8. Bladder cancer.
9. Those taking other antiarrhythmic drugs except beta-blockers.
10. Other diseases cause the patient's life expectancy to be less than 1 year.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2022-11-15 (Estimated); Primary Completion 2024-11-15 (Estimated); Study Completion 2024-11-15 (Estimated)

PRIMARY OUTCOMES:
Number of ICD discharges and mode of electrical therapy (ATP, synchronized cardioversion, electrical defibrillation) | 1 year
  Number of ICD discharges and mode of electrical therapy (ATP, synchronized cardioversion, electrical defibrillation)
Number of ventricular tachycardia/fibrillation events recorded by ICD. | 1 year
  Number of ventricular tachycardia/fibrillation events recorded by ICD.

SECONDARY OUTCOMES:
QRS duration | 1 year
  QRS duration
QT and QTc interval variability | 1 year
  QT and QTc interval variability
QTd | 1 year
  The difference between the longest QT interval and the shortest QT interval in the ECG
Tp-e | 1 year
  Time from T wave apex to T wave end

IPD SHARING:
Plan to Share IPD: No